CLINICAL TRIAL: NCT05192005
Title: Perioperative Blood Pressure and In-hospital Morbidity After Coronary Artery Bypass Surgery
Acronym: PA_PAC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: PA_PAC
Record Dates: First submitted 2021-12-30; First posted 2022-01-14 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Ischemic Cardiopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The prevalence of hypertension is high, estimated at 80% in patients with cardiovascular (CV) disease. The optimal blood pressure (BP) level for CV prevention remains controversial. Data from the literature highlight that the relationship between BP level and mortality is not linear, but rather J-shaped. In particular, in treated hypertensive patients with stable coronary artery disease, a systolic BP below 120 mm Hg is associated with the risk of recurrent coronary events and CV mortality.

An inverse relationship was recently demonstrated between BP level before revascularization procedure and mortality at 3 months and 1 year after the procedure in patients managed for critical ischemia. These data underline the need for a personalized approach to the management of hypertension, especially in elderly hypertensive patients with comorbidities.

The question of the optimal mean BP value also arises in cardiac surgery, especially during extracorporeal circulation in patients undergoing coronary artery bypass grafting. Hypotension during cardiac surgery appears to be associated with renal failure and perioperative mortality in some patients. Conversely, high blood pressure levels (above the cerebral autoregulatory threshold) may be associated with postoperative cognitive impairment and bleeding risk. In hypertensive patients, the autoregulatory capacity of cerebral and renal perfusion is partly impaired, with a greater susceptibility to ischemia in case of hypotension. Personalized blood pressure targets could be beneficial perioperatively with a lower risk of postoperative complications.

The objective of this protocol is to determine a correlation between perioperative mean arterial pressure level and in-hospital morbidity in a population of patients with ischemic heart disease managed for coronary artery bypass grafting (CABG). The results of this descriptive work would make it possible to introduce the problem of the optimal blood pressure target during extracorporeal circulation according to the existence of peripheral arterial damage and preoperative blood pressure values.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age ≥ 18 years
* Patient with ischemic heart disease managed for coronary artery bypass grafting (CABG) between 01/01/2016 and 12/31/2020
* French-speaking patient

Exclusion Criteria:

* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Patient objecting to the use of his data for this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ischemic heart disease managed for coronary artery bypass grafting in the cardiac surgery department at Marie Lannelongue Hospital between 01/01/2016 and 12/31/2020.
Sampling Method: Non-Probability Sample
Enrollment: 1220 (Estimated)
Dates: Start 2023-04-15 (Estimated); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between perioperative mean arterial pressure level in the occurrence of postoperative organ failure | Day 30
  This outcome corresponds to the correlation between preoperative and intraoperative mean arterial pressure levels and the occurrence of postoperative organ failure (composite endpoint).

SECONDARY OUTCOMES:
Correlation between perioperative mean arterial pressure level and occurrence of postoperative organ failure | Day 30
  This outcome corresponds to the correlation between preoperative and intraoperative mean arterial pressure levels and the occurrence of organ failure.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra YANNOUTSOS, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Steg PG, Bhatt DL, Wilson PW, D'Agostino R Sr, Ohman EM, Rother J, Liau CS, Hirsch AT, Mas JL, Ikeda Y, Pencina MJ, Goto S; REACH Registry Investigators. One-year cardiovascular event rates in outpatients with atherothrombosis. JAMA. 2007 Mar 21;297(11):1197-206. doi: 10.1001/jama.297.11.1197. PMID 17374814
- [Background] Bavry AA, Anderson RD, Gong Y, Denardo SJ, Cooper-Dehoff RM, Handberg EM, Pepine CJ. Outcomes Among hypertensive patients with concomitant peripheral and coronary artery disease: findings from the INternational VErapamil-SR/Trandolapril STudy. Hypertension. 2010 Jan;55(1):48-53. doi: 10.1161/HYPERTENSIONAHA.109.142240. Epub 2009 Dec 7. PMID 19996066
- [Background] Vidal-Petiot E, Ford I, Greenlaw N, Ferrari R, Fox KM, Tardif JC, Tendera M, Tavazzi L, Bhatt DL, Steg PG; CLARIFY Investigators. Cardiovascular event rates and mortality according to achieved systolic and diastolic blood pressure in patients with stable coronary artery disease: an international cohort study. Lancet. 2016 Oct 29;388(10056):2142-2152. doi: 10.1016/S0140-6736(16)31326-5. Epub 2016 Aug 30. PMID 27590221
- [Background] Yannoutsos A, Lin F, Billuart O, Buronfosse A, Sacco E, Beaussier H, Mourad JJ, Emmerich J, Lazareth I, Priollet P. Low admission blood pressure as a marker of poor 1-year survival in patients with revascularized critical limb ischemia. J Hypertens. 2021 Aug 1;39(8):1611-1620. doi: 10.1097/HJH.0000000000002821. PMID 33710168
- [Background] Ono M, Arnaoutakis GJ, Fine DM, Brady K, Easley RB, Zheng Y, Brown C, Katz NM, Grams ME, Hogue CW. Blood pressure excursions below the cerebral autoregulation threshold during cardiac surgery are associated with acute kidney injury. Crit Care Med. 2013 Feb;41(2):464-71. doi: 10.1097/CCM.0b013e31826ab3a1. PMID 23263580
- [Background] Ono M, Brady K, Easley RB, Brown C, Kraut M, Gottesman RF, Hogue CW Jr. Duration and magnitude of blood pressure below cerebral autoregulation threshold during cardiopulmonary bypass is associated with major morbidity and operative mortality. J Thorac Cardiovasc Surg. 2014 Jan;147(1):483-9. doi: 10.1016/j.jtcvs.2013.07.069. Epub 2013 Sep 26. PMID 24075467
- [Background] Hori D, Brown C, Ono M, Rappold T, Sieber F, Gottschalk A, Neufeld KJ, Gottesman R, Adachi H, Hogue CW. Arterial pressure above the upper cerebral autoregulation limit during cardiopulmonary bypass is associated with postoperative delirium. Br J Anaesth. 2014 Dec;113(6):1009-17. doi: 10.1093/bja/aeu319. Epub 2014 Sep 25. PMID 25256545